CLINICAL TRIAL: NCT06263868
Title: First Observatory of Precocious and Advanced Puberty in Private Healthcare.
Brief Title: First Observatory of Precocious Puberty.
Acronym: PAPPEL
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1090; 2023-A02313-42 (Other: ID-RCB)
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Puberty, Precocious
Keywords: Early/precocious puberty; advanced puberty; national observatory; private medicine; feasibility
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Precocious puberty group: Girl < 8 years old or boy < 9 years old when the first signs of development appear.
- Advanced puberty group: Girl aged ≥ 8 and < 10 years or boy ≥ 9 and < 11 years old when the first signs of development appear.
- Control group: Boy or girl without any signs of puberty development (Tanner 1)

SUMMARY:
The age of puberty has fluctuated throughout history. Recent data shows an increase in the age of onset of puberty signs, in the United States but also in Europe. A recent Public Health France study published in 2018 reports an increase in the incidence of precocious puberty with geographical heterogeneity. The consequences of these appearances include the early onset of menarche, short adult height and the psychological impact.

Due to a lack of studies and additional data, the reasons for this development are difficult to understand. Among current hypotheses, the entanglement with the evolution of our environment is at the forefront: the action of environmental endocrine disruptors and nutritional factors could play a role in the process of early appearance of pubertal signs.

The establishment of a national observatory for early and advanced puberty in collaboration with pediatric endocrinologists (on the front line) would allow a reliable and precise field approach, capable of supplementing epidemiological data, which are currently insufficient.

The investigators hypothesize that the establishment of an observatory of pubertal advances (early puberty and advanced puberty) in private medicine is possible, with inclusion of at least 75% of eligible patients, and collection of at least 80% of data.

ELIGIBILITY:
Inclusion Criteria:

Precocious puberty group (PP) :

* Suspected precocious puberty (girl aged < 8 years or boy aged < 9 years when the first signs of development* appear)
* Suspected precocious puberty (girl aged < 8 years or boy aged < 9 years when the first signs of development* appear)

Advanced puberty group (AP) :

* Suspected advanced puberty (girl aged ≥ 8 and < 10 years or boy aged ≥ 9 and < 11 years when the first signs of development* appear)
* First consultation with the investigator (pediatric endocrinologist).

Control group :

* Boy or girl without signs of pubertal development (Tanner 1);
* Matched to the PP group on sex and age (+/- 1 year);
* Consultation with the same investigator over the same period (same quarter) as a patient in the PP group

Exclusion Criteria:

All groups

* Consultation with the same investigator over the same period (same quarter) as a patient in the PP group
* Family not speaking French, language barrier.

Max Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients will be recruited in private heathlcare: 2880 patients distributed between the 2 following groups: PP (Precocious puberty group) and PA (Advanced puberty group), and 480 children in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 3360 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2028-06-26 (Estimated)

PRIMARY OUTCOMES:
Number of recruited patients with at least 80% of the main data collected | Up to 48 month
  Number of recruited patients with at least 80% of the main data collected (weight, height, BMI, pubertal stage, date of onset of pubertal signs, questionnaires).
Missing data rate | Up to 48 month
  Missing data rate less than 10% for pubertal stage.
At least 75% of patients included | Up to 48 month
  At least 75% of patients included compared to the number of eligible patients.

CONTACTS AND LOCATIONS:
Overall Officials: Emillie DOYE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (19):
- France (19):
  - Clinique du Val d'Ouest, Écully, Auvergne-Rhône-Alpes
  - Pediatric practice, Lyon, Auvergne-Rhône-Alpes
  - Pediatric practice, Rennes, Brittany Region
  - Pediatric practice, Chambray-lès-Tours, Centre-Val de Loire
  - Pediatric practice, Essey-lès-Nancy, Grand Est
  - Pediatric practice, Levallois-Perret, Hauts-de-Seine
  - Pediatric practice, Fondettes, Indre-et-Loire
  - Polyclinique Bordeaux rive droite, Lormont, Nouvelle-Aquitaine
  - Pediatric practice, Pau, Nouvelle-Aquitaine
  - Pediatric Practice, Pessac, Nouvelle-Aquitaine
  - Clinique rive gauche, Toulouse, Occitanie
  - Pediatric practice, Saint-Nazaire, Pays de la Loire Region
  - Pediatric practice, Aix-en-Provence
  - Hôpital Femme Mère Enfant, Hospices civils de Lyon, Bron
  - Pediatric practice, Marseille
  - Pediatric practice, Nice
  - Clinique Saint jean, Saint-Jean-de-Védas
  - Pediatric practice, Trélazé
  - Pediatric practice, Paris, Île-de-France Region